CLINICAL TRIAL: NCT04887259
Title: A Phase 1 Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Antitumor Activity of LAVA-051 in Patients with Relapsed or Refractory CLL, MM, or AML
Brief Title: Trial of LAVA-051 in Patients with Relapsed/refractory CLL, MM, or AML
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The decision to discontinue LAVA-051clinical trial follows a recent review of the competitive landscape that has continued to evolve (Business decision). The decision is not due to safety concerns.
Sponsor: Lava Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LV2020-001
Record Dates: First submitted 2021-05-03; First posted 2021-05-14 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Chronic Lymphocytic Leukemia; Multiple Myeloma; Acute Myeloid Leukemia
Keywords: CLL; Phase 1 dose escalation; Phase 1 safety; Open label; MM; AML; relapsed; refractory
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Leukemia, Myeloid, Acute; Recurrence | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- LAVA-051 (Experimental): Part 1 (dose escalation): LAVA-051 will be given to patients via intravenous (IV) infusion with dose escalation. A selected group of patients will also receive a low dose of interleukin 2 via subcutaneous injection.
  * Group A: LAVA-051
  * Group B: LAVA-051 + low dose interleukin 2
  Part 2 (dose expansion): patients will receive LAVA-051 at the dose and regimen established in Part 1 of the study
  Interventions: Biological: LAVA-051; Biological: Interleukin 2

INTERVENTIONS:
Biological: LAVA-051 — In part 1 and part 2, LAVA-051 will be administered via intravenous (IV) infusion
Biological: Interleukin 2 — In Part 1 and Part 2, a low dose of interleukin 2 will be given via subcutaneous injection with LAVA-051 in a selected group of patients

SUMMARY:
A phase 1, first-in-human trial to evaluate the safety and tolerability of LAVA-051 in patients with relapsed or refractory Chronic Lymphocytic Leukemia (CLL), Multiple Myeloma (MM), or Acute Myeloid Leukemia (AML).

DETAILED DESCRIPTION:
An open-label, phase 1 dose escalation trial with disease-specific expansion cohorts to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, immunogenicity, and preliminary anti-tumor activity of LAVA-051 in patients with relapsed or refractory CLL, MM, or AML.

The trial was intended to be a Phase 1/2 trial (but the trial never moved forward to Phase 2).

ELIGIBILITY:
KEY INCLUSION CRITERIA

1. Patient must be 18 years of age inclusive or above at the time of signing the informed consent.
2. Patients with documented diagnosis of relapsed or refractory CLL, MM, or AML who have failed to respond to or who have relapsed after prior therapy and are not amenable to standard treatments or for whom no standard treatments are available.
3. Predicated life expectancy of ≥ 3 months.
4. ECOG performance status of 0 or 1.
5. Males or non-pregnant, non-breastfeeding females who are either:

   1. Surgically sterile.
   2. Female of childbearing potential with a negative pregnancy test and compliant with an effective contraceptive regimen.
   3. Female, postmenopausal.
   4. Male compliant with an effective contraceptive regimen.
   5. Male refraining from donating sperm.
6. Capable of giving signed and dated informed consent prior to initiation of any trial-related procedures.

KEY EXCLUSION CRITERIA

1. Prior allogeneic bone marrow transplant if the patient still has active acute or chronic graft versus host disease requiring >10 mg prednisone or equivalent corticosteroids.
2. Concomitant malignancies except carcinoma in situ, basal or squamous cell skin carcinoma. Patients who had no evidence of disease from another primary cancer for 2 or more years are allowed to participate in the trial. Localized non-metastatic prostate cancer, not requiring systemic treatment, and for which no local treatment is planned, is allowed.
3. Uncontrolled or severe intercurrent medical condition.
4. Previous treatment with an aminobisphonsphonate IV (e.g. ibandronate, pamidronate, zoledronate) within 4 weeks prior to initial IMP administration.
5. Known ongoing drug or alcohol abuse in the opinion of the investigator.
6. Previous autologous haematopoietic stem cell transplantation (HSCT) or treatment with Chimeric Antigen Receptor (CAR) T-cell therapy within 6 months prior to initial IMP administration.
7. Immunodeficiency disorders.
8. Patients with Richter's transformation are excluded.

Other eligibility criteria will apply during full screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

PRIMARY OUTCOMES:
Part 1 & Part 2 - Frequency and severity of AEs: | Approximately 6 months
  Frequency, severity, and grading of Adverse Events using the Common Terminology Criteria and grading for Adverse Events (CTCAE) v5.0. CRS will be evaluated using the ASTCT.
Part 1 - Frequency and type of DLT | First 28 days of treatment
  A DLT is defined as an adverse event that is unrelated to disease progression, intercurrent illness, or concomitant medications and is occurring during the first 28 days of treatment. These events will be classified according to the CTCAE v5.0; CRS will be evaluated according to the ASTCT consensus criteria

SECONDARY OUTCOMES:
Part 1 & Part 2: Number of participants with an antitumor response | Approximately 6 months
  Antitumor response for CLL per iwCLL guidelines, MM per IMWG-based response criteria, and AML per ELN criteria
Part 1 & Part 2: Pharmacokinetics of LAVA-051, area under the plasma concentration versus time curve (AUC) | Approximately 6 months
  Area under the plasma concentration versus time curve (AUC) of LAVA-051 will be assessed in all patients treated with LAVA-051
Part 1 & Part 2: Incidence and prevalence anti-LAVA-051 antibodies | Approximately 6 months
  Development of antibodies (anti-drug antibodies) to LAVA-051 will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials Management, Study Director — Lava Therapeutics
Locations (14):
- United States (5):
  - Emory Winship Cancer Institute, Atlanta, Georgia
  - NYU Langone Health, New York, New York
  - Levine Cancer Institute, Atrium Health, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas
- France (2):
  - CHU Lille, Lille
  - University Hospital of Nantes, Nantes
- Netherlands (3):
  - Amsterdam UMC, location VUmc, Amsterdam, North Holland
  - Amsterdam UMC, location AMC, Amsterdam, North Holland
  - Erasmus MC, Rotterdam, South Holland
- Spain (4):
  - University Hospital Vall d'Hebron, Barcelona
  - Cima University of Navarra, Madrid
  - Clinica Universida de Navarra, Pamplona
  - Hospital Clinico Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No